CLINICAL TRIAL: NCT01026805
Title: Retrospective Case Review - Clinical Evaluation of the Interlace Medical 1st Generation Hysteroscopic Morcellator
Brief Title: Clinical Evaluation of the Interlace Medical Hysteroscopic Morcellator
Status: Completed | Type: Observational
Sponsor: Hologic, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: TMP 200901
Record Dates: First submitted 2009-04-30; First posted 2009-12-04 (Estimated); Results first posted 2009-12-04 (Estimated); Last update posted 2012-11-22 (Estimated); Status verified 2012-11

CONDITIONS: Abnormal Uterine Bleeding; Infertility
Keywords: morcellator; hysteroscope; myomectomy; polypectomy; uterine fibroids
MeSH Terms: conditions — Metrorrhagia; Infertility; Leiomyoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hysteroscopic Morcellator: 11 women previously receiving hysteroscopic myomectomy or polypectomy using the hysteroscopic morcellator device.
  Interventions: Device: Interlace Medical 1st Generation Hysteroscopic Morcellator

INTERVENTIONS:
Device: Interlace Medical 1st Generation Hysteroscopic Morcellator — The Interlace Medical hysteroscopic morcellator system has been cleared by the FDA(K073690)and consists of a motor drive unit connected to a 3mm morcellator. The morcellator is approximately 12 cm long and is equipped with an open channel that houses a reciprocating blade. When the motor is activated, the reciprocating blade will cut the tissue within the channel. The tissue travels down the 3mm morcellator shaft cannula via suction coupled to the proximal end of the morcellator and is captured in a tissue trap in a suction canister for pathological diagnosis following the procedure.
  Other Names: MyoSure Tissure Removal System; MyoSure Tissure Removal Device

SUMMARY:
This study assesses the effectiveness of intrauterine fibroid and polyp removal using the Interlace Medical 1st generation hysteroscopic morcellator device based on a retrospective review of medical records of women who have been treated with the device.

DETAILED DESCRIPTION:
A retrospective review of medical records for eleven (11) premenopausal women who had been treated with the new hysteroscopic morcellator was conducted at four hospital or ambulatory surgical center sites. Four physicians performed hysteroscopic operative procedures to remove intrauterine polyps, type 0 (completely within the uterine cavity), type I (mostly within the cavity) and type II (< 40% within the cavity) submucous myomas. Percent pathology removed, total morcellation time, total fluid used, fluid deficit and treatment-related adverse events were assessed. Each of the four treating physicians also evaluated device performance using a 10 point scale (1 = "poor" and 10 = "excellent").

ELIGIBILITY:
Inclusion Criteria:

* female
* at least 18 years old
* treated for intra-uterine submucosal fibroids (Type 0 or 1 myomas and/or polyps using the Interlace 1st generation morcellator device.

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eleven (11) premenopausal women who had been treated with the new hysteroscopic morcellator to resect intrauterine pathology (polyps and submucous myomas).
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2009-02; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Miller, M.D., Principal Investigator — Edward Hospital

RESULTS

PARTICIPANT FLOW:
Recruitment Details: An unselected series of eleven (11) premenopausal women who had been treated with the new hysteroscopic morcellator at four hospital or ambulatory surgical center sites were assessed for this study.
Groups:
- Hysteroscopic Morcellator Treatment Group: Subjects underwent hysteroscopic tissue removal of intrauterine polyps and/or myomas using the Interlace Medical tissue removal device.
Period: Overall Study
Arm/Group | Hysteroscopic Morcellator Treatment Group
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Hysteroscopic Morcellator Treatment Group
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 40.5 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 0
size of fibroid or polyp [Mean (Full Range); unit: mm] — measure size of pathology pre-treament via ultrasound or hysteroscopic exam
  mm | 16.3 [5.0 to 50.0]

OUTCOME MEASURES:

1. Secondary Outcome: Treatment Time Per Patient
Description: mean morcellation(division into and removal of small pieces, as of tissue) time per patient
Time Frame: at time of treatment
Measure: Mean (Full Range); unit: minutes
Arm/Group | Hysteroscopic Morcellator Treatment Group
Number analyzed (Participants) | 11
minutes | 4.3 [0.2 to 22.6]

2. Secondary Outcome: Fluid Volume Per Procedure
Description: mean volume of distension fluid infused into the uterus, per procedure. Distention fluid is used to distend the uterus and provide increased visibility.
Time Frame: at time of treatment
Measure: Mean (Full Range); unit: mL
Arm/Group | Hysteroscopic Morcellator Treatment Group
Number analyzed (Participants) | 11
mL | 5179.0 [600 to 24000]

3. Secondary Outcome: Fluid Deficit Per Procedure
Description: mean fluid deficit per procedure. Fluid deficit is the difference between the amount of fluid which is infused into the patient during the hysteroscopic procedure, and the amount of fluid collected at completion of the procedure.
Time Frame: at time of treatment
Measure: Mean (Full Range); unit: mL
Arm/Group | Hysteroscopic Morcellator Treatment Group
Number analyzed (Participants) | 11
mL | 567.8 [30 to 1900]

4. Secondary Outcome: Resected Tissue Weight Per Patient
Description: mean weight of resected tissue per patient
Time Frame: at time of treatment
Measure: Mean (Full Range); unit: g
Arm/Group | Hysteroscopic Morcellator Treatment Group
Number analyzed (Participants) | 11
g | 10.8 [0.5 to 45.3]

5. Secondary Outcome: Interlace Medical 1st Generation Hysteroscopic Morcellator Cutting Ability - Mean Score
Description: a 10 point scale assessed performance of the Interlace Medical 1st Generation Hysteroscopic Morcellator("1" = "poor" and "10" = "excellent").
Time Frame: 2-3 months post treatment
Population: All treating physicians completed a survey questionnaire.
Measure: Mean (Full Range); unit: scores on a scale
Arm/Group | Hysteroscopic Morcellator Treatment Group
Number analyzed (Participants) | 4
scores on a scale | 9.5 [8 to 10]

6. Secondary Outcome: Adverse Events
Description: Patient medical records were examined to identify any procedure-related or post-treatment adverse events. An adverse event is any undesirable experience (sign, symptom, illness, or other medical event) occurring in a subject, that appears or worsens during a clinical study
Time Frame: 2-3 months post-treatment
Measure: Number; unit: events
Arm/Group | Hysteroscopic Morcellator Treatment Group
Number analyzed (Participants) | 11
events | 0

7. Primary Outcome: Percentage of Tissue Removed
Description: mean percentage of polyp and fibroid tissue removed, as measured on post-treatment hysteroscopic imaging. Images were obtained immediately post treatment, before the subject left the surgical suite.
Time Frame: immediately post-treatment
Measure: Mean (Full Range); unit: Percentage of tissue removed
Arm/Group | Hysteroscopic Morcellator Treatment Group
Number analyzed (Participants) | 11
Percentage of tissue removed | 97.5 [50 to 100]

ADVERSE EVENTS:
Arm/Group | Hysteroscopic Morcellator Treatment Group
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

LIMITATIONS AND CAVEATS:
Small number of cases; retrospective study design

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less